CLINICAL TRIAL: NCT05585346
Title: Photobiomodulation Therapy for Idiopathic Facial Paralysis: Nonrandomized Trial Controlled
Brief Title: Photobiomodulation Therapy for Idiopathic Facial Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBMT-IFP-2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2022-02

CONDITIONS: Bell's Palsy
Keywords: Idiopathic facial paralysis; Bell's palsy; photobiomodulation; RCT
MeSH Terms: conditions — Bell Palsy | interventions — Thiamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture Group (Experimental): LA group used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy). MLS laser is a class IV NIR laser with two synchronized sources (905 nm with 75 W peak power, pulsed mode; 808 nm with power 1 W, continuous mode). Both laser beams were synchronized, the locked waves work with the range 1-2000 Hz.
  In LA group, based on clinical experience, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 7 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST25 (Tian Shu), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong). The acupoints in the limbs and trunk area, were applied bilaterally. Power of laser device is 50%.
  Oral vitamin B1.
  Interventions: Device: MLS laser; Drug: Oral vitamin B1
- Control Group (Active Comparator): LA group used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy). MLS laser is a class IV NIR laser with two synchronized sources (905 nm with 75 W peak power, pulsed mode; 808 nm with power 1 W, continuous mode). Both laser beams were synchronized, the locked waves work with the range 1-2000 Hz.
  In LA group, based on clinical experience, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 7 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST25 (Tian Shu), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong). The acupoints in the limbs and trunk area, were applied bilaterally. Power of laser device is 25%.
  Oral vitamin B1.
  Interventions: Device: MLS laser; Drug: Oral vitamin B1

INTERVENTIONS:
Device: MLS laser — Treatments were performed with MLS laser (Mphi laser, ASA Srl, Italy). MLS laser is a class IV NIR laser with two synchronized sources (laser diodes). The first one is a pulsed laser diode, emitting at 905 nm, with 25 W peak power. The second laser diode (808 nm) was operated in a continuous mode with power 1 W. Both of the laser beams were synchronized, the locked waves work within the range 1-2000 Hz.
Drug: Oral vitamin B1 — Oral vitamin B1 10mg, times/day

SUMMARY:
Objective:

Bell's palsy is characterized by acute, unilateral onset that compromises function and esthetics, exerting a considerable impact on the social, professional, and psychological aspects of the lives of affected individuals. Without treatment, 30% of patients with complete paralysis will not completely recover. Therefore, shortening the recovery time will accelerate the recovery process leading to better results.

The objective of this study was to determine whether photobiomodulation therapy with laser acupuncture therapy could relieve symptoms in patients with Bell's palsy.

Methods:

This study was an open-label, randomized controlled trial including 96 patients that undergoing Bell's palsy. All the patients received oral vitamin B1.

Patients were assigned to the laser acupuncture (LA) group and control group, with 102 patients in each group. LA group were received 4 weeks of Laser treatment (3 times per week), while control group were received sham laser treatment.

Clinical outcome measure comprised the House-Brackmann grading system, Facial Clinimetric Evaluation Scale (FaCE), Sunnybrook facial grading scale (SBFG), and electrophysiological testing, including Electroneuronography (ENoG), Electromyography (EMG) and Blink Reflex. All the measurements were collected at the first day and at the end of study. All reported P values were two-sided and were declared statistically significant when less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of Bell's Palsy. (2) Adults over 18 years of age and under 60 years of age.

Exclusion Criteria:

- (1) Systemic disease, such as severe diabetes, malignant tumors and other serious consumptive diseases.

(2) Serious mental illness or social problems, and neurological disorders. (3) Planning for pregnancy, in pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
The House-Brackmann Facial Nerve Grading System | Change from Baseline number of pathological HB grading at 4-weeks in post-therapy.
  The House-Brackmann facial nerve grading system (HB grading) is based on a 6-grade score that offers a gross evaluation of facial motor function and includes the evaluation of sequelae. The prognoses of patients with House-Brackmann grade I or grade II were considered good, and the prognoses of those with grade 3 or higher were considered poor.
The Sunnybrook Facial Grading System | Change from Baseline scores of SB grading at at 4-weeks in post-therapy.
  The Sunnybrook facial grading system (SB grading) is 13-items, self-reported questionnaire that used to evaluate the facial movement of patients. Among the overall 13 items of question, 3 items are resting symmetry, 5 items are symmetry of voluntary movement, and 5 items are synkinesis. Lower scores of Sunnybrook equate to greater severity of facial paralysis symptoms.

SECONDARY OUTCOMES:
Electroneuronography (ENoG) | Change from Baseline amplitude and potential of CAMP and the numbers of pathological ENoG at at 4-weeks in post-therapy.
  The goal of the Electroneurography (ENoG) testing is to measure the amount of neural degradation that has occurred distal to the site of facial nerve injury by measuring the muscle response to an electrical stimulus. The testing of ENoG involves recording the compound muscle action potential (CAMP) of the mimetic muscles, including Orbicularis oculi, Frontalis muscle, Orbicularis oris and Zygomaticus muscle.
  ENoG is performed first on the healthy side of the face and then on the affected side. Nerve damage or nerve fiber degeneration leads to a decrease or loss of the CAMP. The amplitude of the CAMP on the affected side is compared to the CAMP of the healthy side and expressed as percent (amplitude of the paralyzed side divided by the amplitude of the normal side). A side difference of 30% or bigger is considered pathologic.
Electromyography (EMG) | Change from Baseline amplitude and duration of MUAPs at at 4-weeks in post-therapy.
  EMG is an electrophysiologic measures that indirectly quantify facial nerve function by recording motor unit action potentials (MUAPs) in the muscle of Musculus depressor angulli oris, Frontalis muscle and Orbicularis oris. MUAPs are the spikes in electrical activity generated when a motor unit fires. A motor unit consists of a motor neuron and the corresponding muscle fibers innervated by the neuron.
Blink Reflex | Change from Baseline number of pathological Blink Reflex at 6-months in post-therapy.
  The blink reflex test is to measures the facial nerve since the blink reflex delivers information on facial nerve function with normal trigeminal function. Blink reflex testing involves electrical stimulation of the supraorbital nerve on the affected side combined with a 2-channel simultaneous sEMG recording from both orbicularis oculi muscles. The exit of the supraorbital nerve in the supraorbital foramen is palpated on the rim of the orbit. Stimulation with 10-20 mA and 0.2 ms duration is used to produce a constant reflex.
  In blink reflex testing, two responses, R1 and R2, are analyzed. R1 is the fast ipsilateral response of the orbicularis oculi muscle with a latency of about 10-12 ms. The second bilateral response R2 has a latency of about 30-41 ms.
  The R2 latency differences between both sides higher than 5-8 ms is considered pathologic.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No